CLINICAL TRIAL: NCT04624555
Title: The Utility and Feasibility of Mt-sDNA as a Surveillance Procedure in Colorectal Cancer Survivors
Status: Recruiting | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: CASE14219
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Stage I Colorectal Cancer; Stage II Colorectal Cancer; Stage III Colorectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample for nt-sDNA testing that will be collected within 90 days before their scheduled colonoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research study is to determine whether testing of stool for a panel of markers will enable us to detect polyps and cancer compared to standard testing.

DETAILED DESCRIPTION:
Participants who were diagnosed with Stage I-III colorectal cancer will undergo testing with mt-sDNA followed by a questionnaire about satisfaction with mt-sDNA (multitarget stool DNA panel), prior to their scheduled colonoscopies at years 1 and 4 after diagnosis.

Participants will be asked to provide a stool sample for mt-sDNA (Cologuard) testing that will be collected within 90 days before their scheduled colonoscopy. The kit will be given to the participant by study personnel and mailed back directly to Exact Science.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I, II or III adenocarcinoma of the colon or rectum
* Receipt of preoperative colonoscopy
* Receipt of bowel resection; use of adjuvant chemotherapy or radiation therapy as clinically indicated

Exclusion Criteria:

* Stage IV colorectal cancer
* Surgical treatment with subtotal colectomy or total proctocolectomy
* Diagnosis of inflammatory bowel disease (ulcerative colitis or Crohn's disease)
* Diagnosis of polyposis syndrome including Lynch syndrome or familial polyposis
* Presence of advanced adenomas (1 cm or larger, villous features and/or high grade dysplasia) that were not removed at the preoperative colonoscopy or contained in the resection specimen.
* Inability to provide informed consent
* Inability to understand spoken and written English
* Medical comorbidities that would be contraindications to sedation or that would preclude any benefit of routine surveillance post-resection. These would be at the discretion of the participant's providers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are diagnosed with stage I-III colorectal cancer. All participants who are within 1 year of colon cancer resection will be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of mt-sDNA compared to Colonoscopy | at 1 and 4 years
  Compare the results between mt-sDNA (categorized as a single positive or negative result) with the findings at colonoscopy, the "gold standard". Colonoscopy will be considered positive if an adenoma or carcinoma is found and otherwise negative.
  Sensitivity is defined as True Positive (TP)/(TP+ False Negative (FN))
Specificity of mt-sDNA compared to Colonoscopy | at 1 and 4 years
  Compare the results between mt-sDNA (categorized as a single positive or negative result) with the findings at colonoscopy, the "gold standard". Colonoscopy will be considered positive if an adenoma or carcinoma is found and otherwise negative.
  Specificity is defined as True Negative (TN)/(TN+ False Positive (FP))
Participant acceptance of mt-sDNA as a follow up strategy compared to colonoscopy as measured by the Stool Test Satisfaction Survey. | at 1 and 4 years
  Participant acceptance as measured by the Stool Test Satisfaction Survey, which includes 14 questions scored on a Likert scale. Possible scores ranging from 14 - 70, with higher scores indicating better outcomes.
  Responses will be grouped based on the distribution, but most likely as 1-2 (neutral, unfavorable or least favorable ) versus 3-5 (most favorable or very favorable).

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Cooper, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication
Supporting Information: CSR